CLINICAL TRIAL: NCT01555749
Title: A Randomised, Double-blind, Placebo-controlled, Single Centre, Single Dose Trial, Assessing the Pharmacokinetics of NNC172-2021, Administered Subcutaneously at Two Different Dose Levels, in Healthy Japanese Subjects
Brief Title: Investigation of the Pharmacokinetics of NNC172-2021, at Two Different Dose Levels, in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN7415-3981; 2011-004575-36 (EudraCT Number); U1111-1124-5137 (Other: WHO)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B; Healthy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC172-2021 low dose / Placebo (Experimental)
  Interventions: Drug: NNC172-2021; Drug: placebo
- NNC172-2021 high dose / Placebo (Experimental)
  Interventions: Drug: NNC172-2021; Drug: placebo

INTERVENTIONS:
Drug: NNC172-2021 — One injection administered subcutaneously (s.c., under the skin). Injection of maximum 1.2 mL
Drug: placebo — One injection administered subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetics (how the trial drug is distributed in the body) of NNC172-2021 administered subcutaneously, at two different dose levels, in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese subjects defined as: Subjects born in Japan, time residing outside of Japan does not exceed 5 years, both parents and all 4 grandparents of Japanese descent
* Body weight between 50 and 100 kg, both inclusive
* Body mass index (BMI) between 18.0 and 30.0 kg/m^2, both inclusive

Exclusion Criteria:

* Male subjects who are sexually active and not surgically sterilised who, or whose partner, are unwilling to use two different forms of effective contraception, one of which has to be a barrier method of contraception (e.g. condom with spermicidal foam/gel/film/cream) for the duration of the trial and for 3 months following the last dose of trial medication
* Planned surgery 30 days prior to trial product administration and/or during the entire trial period
* Known hepatic dysfunction during the last 12 months prior to screening (Visit 1)
* Positive urine test for drugs of abuse
* Active hepatitis B and/or hepatitis C infection
* Positive for human immunodeficiency virus (HIV)
* Subjects with clinical signs of thromboembolic events, considered to be at high risk of thromboembolic event or subjects with a known first degree family history of thromboembolism
* Participation in any other trial investigating other products or involving blood sampling within the last 30 days prior to screening
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) such as acetylsalicylic acid (ASA), but not ibuprofen and cyclooxygenase-2 (COX-2) specific inhibitors within 2 weeks prior to trial product administration (Visit 2)
* Positive alcohol test at screening (Visit 1) and/or history of alcohol or drug abuse within the last 12 months prior to screening (Visit 1)
* Smokers; defined as tobacco users smoking more than 5 cigarettes per day or the corresponding amount of tobacco consumption
* Blood donation within the last 3 months prior to screening and/or during the entire trial period
* Strenuous exercise (as judged by the trial physician) within the last 4 days prior to screening (Visit 1)

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-03-12 (Actual); Primary Completion 2012-05-08 (Actual); Study Completion 2012-05-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time point 0 to infinity (AUC0-∞) of NNC172-2021 | Week 5

SECONDARY OUTCOMES:
Maximal concentration of NNC172-2021 (Cmax) | Week 5
Time point for maximal concentration (tmax) | Week 5
Terminal half-life (t1/2) | Week 5
Number of adverse events (AEs) | Week 5
Presence of antibodies against NNC172-2021 | Week 5
Residual tissue factor pathway inhibitor (TFPI) functionality measured by coagulation factor Xa (FXa) generation | Week 5
TFPI concentration measured by tissue factor pathway inhibitor (TFPI) enzyme-linked immunosorbent assay (ELISA) | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com